CLINICAL TRIAL: NCT03523624
Title: Factor XIII and Other Biomarkers in ST Segment Elevation Myocardial Infarction
Acronym: eXIST
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Vittorio Pengo, Associate Professor of Cardiology, University of Padova
Other Study IDs: eXIST-DCTV
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Factor XIII Deficiency; ST-Elevation Myocardial Infarction; Myocardial Haemorrhage; Coronary Microvascular Disease
Keywords: factor XIII; intramyocardial haemorrhage; microvascular injury; STEMI; cardiac magnetic resonance
MeSH Terms: conditions — Factor XIII Deficiency; ST Elevation Myocardial Infarction; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma will be stocked for FXIII determination
Oversight: Data Monitoring Committee: No

SUMMARY:
In medical practice, a combination of clinical exam, electrocardiograms, circulating biomarkers, and imaging is used to gain insights on the prognosis after myocardial infarction. Novel molecular non-invasive tools are needed that help clinicians overcome the adverse events of post-myocardial infarction remodelling and thereby achieve improved therapy for its prevention.

Coagulation factor XIII (FXIII) decay has been linked to major adverse cardiac events (MACE) in patients with acute coronary syndromes. Given the correlation between both intramyocardial haemorrhage and microvascular damage with acute phase complications in ST-elevation myocardial infarction, we hypothesise that excessive FXIII decay within the first week may predict acute phase outcomes in these patients. If this holds true, FXIII determination could be used as diagnostic and prognostic tool.

DETAILED DESCRIPTION:
Background:

The reduction of mortality in acute myocardial infarction (AMI) is achieved by the efficacy of the current therapeutic strategies focused on an early reopening of the culprit coronary artery, by either medical or mechanical reperfusion. Primary percutaneous coronary intervention (PCI) represents the most effective way to limit infarct size and reduce transmural extension of necrosis. Although coronary artery recanalization represents the most effective way to reduce infarct size, the process of reperfusion may itself produce a series of consequences including intramyocardial haemorrhage (IMH) and microvascular injury (MVO) contributing to the 'no reflow' phenomenon. MVO is an early event followed by intramyocardial haemorrhage that plays a role later in reperfusion injury. Both luminal obstruction (microvascular damage by neutrophil plugging, platelets and emboli) and external compression (by oedema and haemorrhage) are allegedly linked with no-reflow, however, the real mechanism underlying this complex time-sensitive phenomenon remains to be fully understood. MVO and IMH in ST-elevation myocardial infarction are independent predictor of adverse left ventricle remodelling, independently of the initial infarct size, and predict MACE.

The diagnosis of no-reflow is usually made when post-procedural thrombolysis in myocardial infarction (TIMI) flow is <3, or in the case of a TIMI flow of 3 when myocardial blush grade is 0 or 1, or when ST resolution within 4 h of the procedure is <70%. It can be assessed using cardiac magnetic resonance (CMR) techniques, where they appear as dark zones on delayed post-contrast sequences or contrast echocardiography.

FXIII is a protransglutaminase that becomes activated by thrombin and catalyses the formation of crosslinked fibrin mesh in the final stage of the clotting cascade. Blood coagulation FXIII is thought to play a role in wound healing and tissue repair. FXIII is present in plasma, platelets, monocytes, and macrophages, all of which are involved in infarct healing. In an experimental model, mice lacking FXIII suffer from impaired wound healing and fatal rupture of the left ventricle after myocardial infarction. This phenomenon was observed in 100% of homozygous and, interestingly, in 100% of the heterozygous FXIII-knockout mice, despite a FXIII plasma level of 70%. Replenishment of FXIII during the 5-day acute and subacute period of infarct healing restored survival rates of FXIII-deficient mice to that of wild-type mice. In addition, reduced FXIII activity imaged via single photon emission computed tomography predicted adverse infarct healing after MI in mice. In contrast, increased intracardiac FXIII activity via induction of high FXIII zymogen plasma levels improved cardiac healing. Moreover, FXIII levels were significantly diminished in myocardial biopsies of human ruptured MI. In a case series of 25 patients with acute MI, a mean decrease of initially normal FXIII plasma values by 25% was reported during the first week after the ischemic event. During the first week after MI, an acute phase reduction in FXIII plasma levels has been described, with the nadir of reduction on day 3-6 after the acute event.

FXIII thus seems to mediate the formation of a well-cemented scar, reducing MVO and IMH and improve healing and left ventricle remodelling.

Aim of the study:

We will perform a prospective observational study to identify how the differences in FXIII levels in ST-elevation myocardial infarction patients relate with intramyocardial haemorrhage and microvascular damage as detected by cardiac magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* patients with the clinical presentation of ST-elevation myocardial infarction within 12 h of symptom onset and with persistent ST-segment elevation or new or presumed new left bundle branch block and undergoing primary percutaneous coronary intervention (PCI)

Exclusion Criteria:

* patients with late presentation ST-elevation myocardial infarction (beyond the first 12h after onset of symptoms) or ineligible for mechanical reperfusion therapy
* contraindications to cardiac magnetic resonance
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that present in the Padova University Hospital Coronary Care Unit with a ST-elevation myocardial infarction will be screened
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
FXIII decay correlation with intramyocardial haemorrhage/microvascular damage | average of 6 days
  FXIII decay will be correlated with intramyocardial haemorrhage/microvascular damage as assessed by cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padua, Cardiology Clinic, Padua, PD, Italy